CLINICAL TRIAL: NCT02469740
Title: Peripheral Endothelial Function Assessment of Patients on Ticagrelor vs. Clopidogrel Who Have Undergone Percutaneous Coronary Intervention - a Randomised, Crossover Study.
Brief Title: Peripheral Endothelial Function Assessment of Patients on Ticagrelor vs. Clopidogrel Who Have Undergone PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Ronstan Lobo, MB, BCh, BAO (Hons), BMedSc (Hons), MRCPI, MRCP(UK), University Hospital of Limerick
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RON004; 2015-000334-30 (EudraCT Number)
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Myocardial Ischemia; Coronary Artery Disease; Endothelial Dysfunction
Keywords: Ticagrelor; Clopidogrel; Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Patients in this group will be prescribed ticagrelor 90 mg BD for 4 weeks.
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Patients in this group will be prescribed clopidogrel 75 mg OD for 4 weeks
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Patients that are randomly selected to receive ticagrelor during the first phase of the study will receive the dose of 90 mg BD orally. This will be continued for 4 weeks before the endothelial function test will be performed. If the patients are assigned in the 2nd phase of the study, they will receive 90 mg BD orally for 5 weeks (4 weeks plus a 1 week washout period).
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Clopidogrel — Patients that are randomly selected to receive ticagrelor during the first phase of the study will receive the dose of 75 mg OD orally. This will be continued for 4 weeks before the endothelial function test will be performed. If the patients are assigned in the 2nd phase of the study, they will receive 75 mg OD orally for 5 weeks (4 weeks plus a 1 week washout period).
  Other Names: Plavix, Clodel
  Arms: Clopidogrel

SUMMARY:
Usage of antiplatelet agents and cardiac procedures such as coronary angioplasty has dramatically improved the morbidity and mortality associated with coronary artery disease. In patients with a coronary stent, dual antiplatelet therapy is recommended. Aspirin is the main antiplatelet agent used. For many years, clopidogrel was the second antiplatelet of choice. Recent studies have revealed new antiplatelet drugs that can substitute clopidogrel, one of which is ticagrelor. The degree to which ticagrelor reduced the overall mortality compared to clopidogrel in the PLATO trial suggested that ticagrelor possibly has a pleiotropic effect and that the reduction in mortality is not simply due to its antiplatelet effects. The ticagrelor molecule resembles adenosine. Adenosine has been shown to be cardioprotective.

The aim of this project is to study the effects of ticagrelor on the arterial system using a noninvasive method. The study will employ the measurement of peripheral endothelial function of patients who undergo percutaneous coronary intervention who are on ticagrelor vs. clopidogrel using a cross over trial design.

DETAILED DESCRIPTION:
Cardiovascular disease remains the most common cause of death in Ireland. Usage of antiplatelet agents and cardiac procedures such as coronary angioplasty has dramatically improved the morbidity and mortality associated with coronary artery disease. In patients with a coronary stent, dual antiplatelet therapy is recommended. Aspirin is the main antiplatelet agent used. For many years, clopidogrel was the second antiplatelet of choice. Recent studies have revealed new antiplatelet drugs that can substitute clopidogrel, one of which is ticagrelor. Ticagrelor received approval from regulatory authorities such as the Food and Drug Administration and the European Medicines Agency based on the PLATO trial which demonstrated a reduction in overall mortality and thrombotic cardiovascular events when compared to clopidogrel. Ticagrelor is approved in Europe and specifically in Ireland for use in patients with ACS and in patients undergoing coronary angioplasty. The degree to which ticagrelor reduced the overall mortality compared to clopidogrel in the PLATO trial suggested that ticagrelor possibly has a pleiotropic effect and that the reduction in mortality is not simply due to its antiplatelet effects. The ticagrelor molecule resembles adenosine. It has been shown that ticagrelor increases adenosine concentration, by interfering with its red blood cells' uptake and by inducing the release of ATP which is then converted to adenosine. Adenosine has been shown to be cardioprotective.

Peripheral Arterial Tonometry (EndoPAT 2000 system (Itamar Medical, Caesarea, Israel) is a method for evaluating endothelial dysfunction. The device has received a CE mark (approved for use in Europe). It uses a non-invasive assessment called fingertip pulse amplitude tonometry.

The reactive hyperaemia response as detected by the reactive hyperaemia index (RHI) has been shown to be related to multiple traditional and metabolic risk factors. It has also been found to positively correlate with flow mediated dilatation (FMD) and coronary vasoreactivity as assessed by intracoronary acetylcholine. A significant advantage of the endoPAT device is the reproducibility of results when compared to FMD in assessment of peripheral endothelial function. Smaller studies have shown positive effects of ticagrelor on endothelial function assessment compared with clopidogrel or prasugrel but no randomised study has been done to date.

The aim of this project is to study the effects of ticagrelor on the arterial system using a noninvasive method. The study will employ the measurement of peripheral endothelial function of patients who undergo percutaneous coronary intervention who are on ticagrelor vs. clopidogrel using a cross over trial design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol
* Subjects must be male or female, aged 18 years or above at baseline
* Diagnosed with coronary artery disease and undergone PCI
* Female subjects of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 12 months (as per guidelines on patients undergoing PCI who are on antiplatelet therapy).
* Female subjects' urine pregnancy test performed at the baseline visit must be negative (which is required by local hospital policy in order to undergo PCI).

Exclusion Criteria:

* Allergy/hypersensitivity to study medications or their ingredients
* Contraindications to either clopidogrel or ticagrelor:

  * Ticagrelor contraindications - active bleeding, history of intracranial haemorrhage, moderate to severe hepatic impairment, dialysis, uric acid nephropathy, co-administration of a strong CYP3A4 inhibitor (e.g. ketoconazole, clarithromycin, nefazodone, ritonavir and atazanavir), history of sick sinus syndrome or high degree AV block without pacemaker protection
  * Clopidogrel contraindications - severe hepatic impairment, active bleeding
* On treatment with oral anticoagulant (vitamin K antagonist, dabigatran, rivaroxaban, apixaban)
* Unable to follow up in research centre (for example, due to logistic difficulties)
* Female subjects who are pregnant or breast-feeding, or considering becoming pregnant during the study.
* Subjects who have participated in another study and received any other investigational agent within the previous 12 months
* Subjects unable to provide written informed consent within 24 hours of PCI (for example, intubated patients)
* Subjects who have a history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Use of both left and right radial access for PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with endothelial dysfunction (Reactive Hyperemia index of < 1.67 using the non-invasive Endo-PAT 2000 device) on ticagrelor versus clopidogrel. | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kiernan, Study Chair — University Hospital of Limerick
Locations (1):
- University Hospital Limerick, Dooradoyle, Limerick, Ireland